CLINICAL TRIAL: NCT06584695
Title: Analgesic Efficacy of External Oblique Intercostal Block Versus Subcostal Transversus Abdominis Plane Block in Open Surgical Nephrectomy
Brief Title: Analgesic Efficacy of External Oblique Intercostal Block vs Subcostal Transversus Abdominis Plane Block in Open Surgical Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelbaset Mostafa, Specialist of Anesthesia, Surgical Intensive Care & Pain Relief, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2407-201-013
Record Dates: First submitted 2024-08-31; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Analgesic Efficacy; External Oblique Intercostal Block; Subcostal Transversus Abdominis Plane Block; Open; Nephrectomy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transversus abdominis plane group (Experimental): patients will receive unilateral ultrasound-guided oblique subcostal transversus abdominis plane block block
  Interventions: Drug: Transversus abdominis plane block
- External oblique intercostal group (Experimental): Patients will receive unilateral ultrasound-guided external oblique intercostal block
  Interventions: Drug: External Oblique Intercostal Plane Block
- Control group (Active Comparator): Patients will receive IV morphine 0.1mg/kg after induction of general anesthesia.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Transversus abdominis plane block — Patients will receive transversus abdominis plane block with an oblique subcostal approach in the supine position. The anesthesiologist will place the linear ultrasound transducer obliquely on the upper abdominal wall along the subcostal margin near the xiphisternum of the sternum in the midline of the abdomen. The anesthesiologist will direct a 22G, 80 mm needle toward the transversus abdominis fascia and inject 25 mL of 0.25% bupivacaine between the rectus abdominis and transversus abdominis muscles along the subcostal line.
  Arms: Transversus abdominis plane group
Drug: External Oblique Intercostal Plane Block — Patients will receive external oblique intercostal block the patient will be in the supine position with their ipsilateral arm abducted, A linear ultrasound transducer will be placed in the sagittal plane between the midclavicular and anterior axillary lines at the level of sixth rib, with the orientation marker directed cranially. The skin will be sterilized, and the probe will be placed over the sixth rib medial to the anterior axillary line in a parasagittal orientation the in-plane technique with a 22G, 80 mm block needle will be used to inject 25 ml of 0.25% bupivacaine into the external oblique intercostal plane.
  Arms: External oblique intercostal group
Drug: Control group — Patients will receive IV morphine 0.1mg/kg after induction of general anesthesia.
  General anesthesia induction will be performed with fentanyl 1-2 μg/kg, propofol 2-3 mg/kg, and rocuronium 0.6 mg/kg and maintained with sevoflurane.
  Arms: Control group

SUMMARY:
To compare the efficacy of unilateral ultrasound-guided oblique subcostal transversus abdominis plane block with unilateral ultrasound-guided external oblique intercostal plane block in providing intraoperative and postoperative analgesia in cancer patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
Open surgery remains one of the procedures used for those patients requiring partial or radical nephrectomy and is associated with a high incidence of severe immediate postoperative pain and chronic pain the months following surgery.

Regional anesthesia techniques are frequently recommended for pain control in open nephrectomy as they decrease the need for parenteral opioid and improve patient satisfaction.

Although abdominal wall blocks are known to decrease opioid requirements without causing epidural associated hypotension, their role in flank surgeries has been less well-established. The dermatomes that need to be covered in flank incision are T9 to T11.

Studies have confirmed that ultrasound-guided (USG) transversus abdominis plane (TAP) block is an effective method of analgesia for upper abdominal surgeries, lower abdominal surgeries and kidney transplantation with minimal side effects.

The external oblique intercostal (EOI) block is a novel method providing simple and effective somatic analgesia to the upper abdomen with minimal side effects. Other advantages include easy sonoanatomy (even in obese patients), being performed in the supine position, and no anticoagulation concern

ELIGIBILITY:
Inclusion Criteria:

* Age (18-65) year.
* Both sexes.
* American Society of Anesthesiologists (ASA) class II and III.
* Cancer patients candidate for open nephrectomy .

Exclusion Criteria:

* Patient refusal.
* Skin lesions or infection at the site of proposed needle insertion.
* Cognitive disorders.
* History of psychiatric disorders or drug abuse.
* Patients allergic to medication used.
* ASA class IV.
* Coagulopathy.
* Body mass index (BMI) more than 35.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours after surgery
  Degree of pain by Numerical rating scale (NRS)score. NRS (0 pain represents "no pain" while 10 pain represents "the worst pain imaginable"). scores will be registered at rest and movement immediately after surgery and at two, six, 12 and 24 hours after surgery, when the (NRS) was > 4, IV morphine PCA will be initiated with continuous rate of 1 mg/hr, a patient demand bolus of 1mg and with lockout time of 10 minutes based on the patient weight and gender. the first time to the rescue analgesia needed and the top up doses will be recorded.

SECONDARY OUTCOMES:
Mean arterial pressure | Till the end of surgery (up to 2hours)
  Mean arterial pressure will be recorded intraoperative till the end of surgery.
Heart rate | Till the end of surgery (up to 2hours)
  Heart rate will be recorded intraoperative till the end of surgery.
Opioids consumption | 24 hours after surgery
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 pain represents "no pain" while 10 pain represents "the worst pain imaginable"). when the (NRS) was > 4, IV morphine PCA will be initiated with continuous rate of 1 mg/hr, a patient demand bolus of 1mg and with lockout time of 10 minutes based on the patient weight and gender. the first time to the rescue analgesia needed and the top up doses will be recorded.
Morphine consumption | 24 hours after surgery.
  When the numeric rating scale (NRS) was >4, IV morphine PCA will be initiated with continuous rate of 1 mg/hr, a patient demand bolus of 1mg and with lockout time of 10 minutes based on the patient weight and gender. the first time to the rescue analgesia needed and the top up doses will be recorded.
  Each patient will be instructed about postoperative pain assessment with the NRS score. NRS (0 pain represents "no pain" while 10 pain represents "the worst pain imaginable").NRS will be registered at rest and movement immediately after surgery and at two, six, 12 and 24 hours after surgery.
Time to rescue analgesia. | 24 hours after surgery
  Time to rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Incidence of complications | 24 hours after surgery
  Incidence of complications will be recorded such as pneumothorax, local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.